CLINICAL TRIAL: NCT02368275
Title: Role of Genetic, Neurophysiological and Psychological Factors in the Development of Postsurgical Neuropathic Pain After Breast Surgery for Cancer
Brief Title: Genetic, Neurophysiological and Psychological Risk Factors for Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Hospital Ambroise Paré Paris (Other)
Collaborators: Hopital Foch (Other)
Responsible Party: Principal Investigator, Nadine ATTAL, Principal investigator, Hospital Ambroise Paré Paris
Other Study IDs: Predictive cohort
Record Dates: First submitted 2015-02-13; First posted 2015-02-23 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples will use GWAS to detect potential genetic risk factors for neuropathic pain. These data will be analysed in Oxford laboratory (McCarthy).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- prospective cohort of patients undergoing mastectomy: Prospective cohort
- cross sectional cohort of patients: Cross sectional cohort

SUMMARY:
The objective of these cohorts is to detect potential genetic, neurophysiological psychological and cognitive risk factors for the development of chronic postsurgical pain including neuropathic pain.

DETAILED DESCRIPTION:
This new study will enroll patients undergoing mastectomy or thoracotomy for cancer. They will be three cohorts :

* one prospective cohort constituted of women undergoing breast surgery in René Huguenin Hospital (Saint Cloud) and followed for up to one year after surgery.
* another cross sectional cohort constituted of patient association (Seintinelle) including women operated up to 2 years previously from breast surgery.
* One prospective cohort constituted of women or men undergoing thoracotomy in Foch hospital (Suresnes) and followed for up to one year after surgery.

The main objectives of these cohorts will be to detect potential genetic, neurophysiological, psychological and cognitive risk factors for the development of chronic postsurgical neuropathic pain.

These patients will questioned about demographics, age, sex, body mass index. A large neuropsychological and psychological battery of tests will be conducted. Sensory function will assessed using quantitative sensory testing. Biological samples will analyse potential genetic factors in the development of neuropathic pain after surgery. Conditioned pain modulation, threshold tracking and quantitative sensory testing will also be assessed in subgroup of patients.

The prospective cohort will be assessed before surgery then 3, 6 and 12 months after surgery. The cross sectional cohort will be assessed during one to two visits in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for breast cancer or thoracotomy for lung cancer followed during the course of the study or patients from the French cohort Seintinelle already operated from breast surgery over the past 2 years.

Exclusion criteria :

* Patients are not included if they have clinically significant or unstable psychiatric or somatic conditions (e.g. major depression, psychosis, uncontrolled diabetes mellitus or hypertension, neurological disorders, immune disease, body mass index > 45), past or present substance abuse or any cognitive deterioration based on past medical history, semi-structured interview and lack of completion or full understanding of questionnaires.
* Bilateral mastectomy (for women undergoing breast surgery)
* Presence of pain before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first group of patients consists of women recruited from René Huguenin Hospital (Saint Cloud, Ile de France) for mastectomy or lumpectomy to treat breast cancer, with axillary lymph node dissection in all cases.
  The second cohort will consist of women already operared of breast surgery in the last 2 years.
  The third cohort will consist of men or women recruited from Foch hospital (Suresnes, Ile de France) for thoracotomy for cancer.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
neuropathic pain | 3, 6 and 12 months after surgery in the prospective cohort
  neuropathic pain assessed with the DN4 questionnaire

SECONDARY OUTCOMES:
chronic postsurgical pain | 3, 6 and 12 months after surgery
  chronic pain questionnaire identification

CONTACTS AND LOCATIONS:
Overall Officials: Nadine ATTAL, MD, PhD, Principal Investigator — Principal Investigator
Locations (2):
- France (2):
  - Hôpital Foch, Suresnes, Hauts De Seine
  - Hôpital Ambroise Paré, Boulogne-Billancourt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sperandio G, Baudic S, Bennedsgaard K, Grosen K, Andersen IS, Finnerup NB, Albi-Feldzer A, Flor H, Nees F, Bouhassira D, Attal N. Somatic and psychological predictors of chronic postsurgical pain in cancer patients: a machine learning approach in a longitudinal two-centre study. Br J Anaesth. 2026 Jan 7:S0007-0912(25)00847-5. doi: 10.1016/j.bja.2025.12.002. Online ahead of print. PMID 41506969